CLINICAL TRIAL: NCT06338280
Title: Remote Observed Methadone Evaluation Phase II (ROME II): Retention and Costs of Care
Brief Title: Remotely Observed Methadone Evaluation II
Acronym: ROME II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sonara Health (Industry)
Collaborators: Chestnut Health Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VDW002
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sonara-enabled (Experimental)
  Interventions: Other: Sonara
- Treatment as usual (No Intervention)

INTERVENTIONS:
Other: Sonara — Sonara virtual dosing window and engagement platform
  Arms: Sonara-enabled

SUMMARY:
Methadone is an effective treatment for severe opioid use disorder (OUD), but access is limited due to the requirement of daily observed dosing by most opioid treatment programs (OTPs). Sonara Health designed a HIPAA-compliant web-application called Sonara that features integrated video dosing recording, a tamper-evident seal, and an innovative measurement-based care (MBC) framework called the Opioid Craving Visual Analogue Scale (OC-VAS) to facilitate methadone take-homes while providing evidence of appropriate use and monitoring patient outcomes. Phase II of this SBIR aims to compare Sonara against usual take-homes to assess its impact on retention in care, opioid use, patient outcomes, and costs of care.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in a randomized trial
* Able to complete study instruments and interviews

Exclusion criteria:

* Less than 18 years of age
* Pregnant or planning to be pregnant
* Currently involved in the criminal justice system
* Serious mental health problems
* Treated with buprenorphine

Please note: The enrollment target (2.5 randomizations per week over 50 weeks) includes oversampling women and under-represented racial/ethnicity groups (i.e., at least 10 or more individuals per group who identify as Black, Hispanic, and American Indian/Alaskan Native).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Retention | 24 weeks
  Length of time the patient remains in treatment after study enrollment
Take homes received over time | 24 weeks
  The number of take home doses of methadone received at 4-, 12-, and 24-weeks following randomization

SECONDARY OUTCOMES:
Opioid cravings | 24 weeks
  Opioid craving visual analog scale (OC-VAS), a single-item, patient-reported outcome measure that captures the severity of cravings, reported on a 0-100 scale
Urine toxicology | 24 weeks
  A qualitative test that detects the presence of commonly used illicit substances or their metabolites in a urine sample
Opioid withdrawal severity | 24 weeks
  Subjective Opioid Withdrawal Scale (SOWS) - a self-administered scale for grading opioid withdrawal symptoms. It contains 16 symptoms whose intensity the patient rates on a scale of 0 (not at all) to 4 (extremely)
Health-related quality of life | 24 weeks
  CDC (Health-related quality of life) HRQOL-14 "Healthy Days Measure" - 14-item questionnaire that assesses an individual's perceived physical and mental health status over the past 30 days, including self-rated health, recent days of poor physical or mental health, and activity limitations
Drug Abuse Treatment Costs Analysis | 24 weeks
  A standardized method for estimating the economic costs of substance abuse treatment programs, including both direct costs (such as personnel, supplies, and facilities) and indirect costs (such as overhead and administrative expenses)

CONTACTS AND LOCATIONS:
Locations (1):
- FGC Wabash, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No